CLINICAL TRIAL: NCT03163381
Title: Apatinib Second Line Treatment for Advanced Osteosarcoma and Soft Tissue Sarcomas ,Openting ,Single Center, One-armed Clinical Study.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Principal Investigator, YaoWeitao, Deputy Director, Henan Cancer Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AHEAD-HNP007
Record Dates: First submitted 2017-05-18; First posted 2017-05-23 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Osteosarcoma, Advanced
Keywords: first-line treatment failure; one measurable lesion
MeSH Terms: conditions — Osteosarcoma | interventions — apatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib (Experimental): Apatinib 500mg/d from day 1 to day 28, repeated every 28 days until progressive Disease(PD) .
  Interventions: Drug: Apatinib

INTERVENTIONS:
Drug: Apatinib — Apatinib 500mg,po,qd,medicine to disease progression.

SUMMARY:
Apatinib second line treatment for Advanced osteosarcoma and soft tissue sarcomas ,openting ,single center, one-armed clinical study.

DETAILED DESCRIPTION:
The treatment of bone and soft tissue sarcomas are usually surgery and chemotherapy,advanced cases cannot be removed through surgical method for multiple metastasis,advanced cases Most advanced cases with chemotherapy is given priority to, but the effect is not ideal.Apatinib main through inhibit VEGFR to give play to Anti-angiogenesis effect to treatment of malignant tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Subject joined the study of his or her own free will , signed informed consent;
2. Subject that diagnosed with advanced osteosarcoma by pathology and first-line treatment failure, at least have one measurable lesion ; Or confirmed by the pathology of advanced soft tissue sarcomas, at least have one measurable lesion,main include Synovial sarcoma、 Leiomyosarcoma、Alveolar soft part sarcoma、Undifferentiated pleomorphic sarcoma/malignant fibrous histiocytoma、Adipocytic Tumors、 Fibrosarcoma、Clear cell sarcoma、Epithelioid sarcoma、Malignant peripheral nerve sheath tumor、Undifferentiatedsarcoma、 Rhabdomyosarcoma、chondrosarcoma、Osteosarcoma、Dermato- fibrosarcoma protuberans、GIST、Primitiveneuroectodermal tumor、Inflammatory myofibroblastic tumor、Malignant mesothelioma； 3）Within the past 6 months, Subject using at least one chemotherapy regimens (including anthracycline-based) failured (except gland alveolar soft tissue sarcoma); 4）18 to 70 years (including 18 and 70 ), men and women there is no limited. 5）ECOG PS score: 0 ~ 1; 6）Estimated survival period more than 3 months; 7）Main organs function within 7 days before the treatment, meet the following criteria:

   1. Blood routine examination standard( without blood transfusion condition in 14 days) :HB≥90g/L;②ANC≥1.5×109/L;③PLT≥80×109/L
   2. Blood biochemical examination must meet the following criteria:

      ① TBIL≤1.5ULN ；②ALT and AST≤2.5ULN，if With hepatic metastatic carcinoma，ALT and AST≤5ULN；③Cr≤1.5ULN或CCr≥60ml/min；
   3. Doppler ultrasound assessment: LVEF normal or low limit (50%).

      Exclusion Criteria:

      - 1）Subject with hypertension, and after antihypertensive drug therapy can't to the normal range (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg), Ⅱ or higher level of coronary heart disease, arrhythmia (include QTc prolonging, male > 450 ms, female > 470 ms) and cardiac insufficiency; 2）Subject used targeted therapy of vascular endothelial growth inhibitor drug previous, include Sunitinib, Sorafenib ,bevacizumab, imatinib and so on.

      3）With other malignant tumor before or at the same time, but except the cured skin basal cell carcinoma and carcinoma in situ of cervix.

      4）Subject accepted anticancer therapy before with NCI CTCAE classification > 1 grade toxicity reaction.

      5）Has multi-factors that effect of oral drug absorption(, such as unable to swallow, nausea or vomiting, chronic diarrhea and intestinal obstruction, etc.); 6）Special note: subject with gastrointestinal bleeding risk can't enrolled the study, include: (1) there are active peptic ulcer lesions, and defecate occult blood (+ +);(2)Subject with medical history include Melena、hematemesis in three months;(3) Subject must be of gastroscopy with defecate occult blood, clear whether deposit organic gastrointestinal tract diseases; 7）Subject with coagulant function abnormality (INR > 1.5 x ULN, APTT > 1.5 x ULN), bleeding tendency; 8）Didn't heal wounds for a long time or fracture. 9）Subject with active bleeding or within 30 days after Major surgery. 10）Intracranial metastasis; 11）Pregnant or lactating women; 12）cell toxic drug therapy, radiation therapy 3 weeks after treatment; Once took two or more targeted drugs, or once took other targeted drugs 3 months before enrollment.

      13）Suffered from other malignant tumor for the past three years. 14）Investigator considered that there may be exist any situation that can damage subject or result in subject can't meet or carry out Investigator requests.

      15）huge transfer/recurrent lesions(tumor size greater than 5 cm). 16）malignant pleuraleffusion or peritoneal effusion, caused NCI CTCAE grading more than 2 levels of breathing difficulties; Description: oversized tumor load often indicates poor blood supply, lead to drug unable to effectively into the tumor, in order to accurately assess the treatment effects apatinib to the soft tissue sarcomas, Our study do not accept with huge transfer recurrent focal (tumor diameter greater than 5 cm) of the patients into groups temporarily .

      17）Allergy to any ingredient about apatinibshould be ruled out; 18）Subject with severe liver and renal failure (level 4) should be ruled out; 19）Subject has a history of psychiatric drugs abuse and can't quit or have a mental disorder; 20）According to the investigator's judgment, subject who has concomitant diseases that serious to endanger the safety or impact subject to complete the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — 18 to 70 years (including 18 and 70 ).
Enrollment: 40 (Estimated)
Dates: Start 2017-04-11 (Actual); Primary Completion 2017-10-11 (Estimated); Study Completion 2019-04-11 (Estimated)

PRIMARY OUTCOMES:
progress free survival | 6 months
  time from study drug treatment to tumor progress

SECONDARY OUTCOMES:
overall survival | up to 24 months
  Time from study drug treatment to die

CONTACTS AND LOCATIONS:
Locations (1):
- Henan cancer hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided
Temporarily not sure whether to be Shared the data.

REFERENCES:
- [Derived] Hattinger CM, Patrizio MP, Magagnoli F, Luppi S, Serra M. An update on emerging drugs in osteosarcoma: towards tailored therapies? Expert Opin Emerg Drugs. 2019 Sep;24(3):153-171. doi: 10.1080/14728214.2019.1654455. Epub 2019 Aug 14. PMID 31401903